CLINICAL TRIAL: NCT02593630
Title: Field Study of Unicirc Circumcision in Adolescent Boys, Aged 12 to 15 Years.
Brief Title: Unicirc Adolescent 12-15 Year Old Boys
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Simunye Primary Health Care (Other)
Responsible Party: Principal Investigator, Peter Millard, PI, University of New England
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Unicirc Adolescent
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unicirc circumcision (Experimental): Unicirc circumcision under topical anaesthetic, wound sealing with cyanoacrylate tissue adhesive
  Interventions: Device: Unicirc circumcision

INTERVENTIONS:
Device: Unicirc circumcision — Unicirc circumcision under topical (EMLA) anaesthesia, wound sealing with cyanoacrylate tissue adhesive

SUMMARY:
This is a field case series of Unicirc under topical anaesthetic among adolescent boys, aged 12 to 15 years.

DETAILED DESCRIPTION:
Boys are healthy, without severe anatomic abnormalities complicating circumcision. Boys with moderate phimosis and tight frenulum were included. Informed assent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* healthy boys desiring circumcision

Exclusion Criteria:

* current illness
* bleeding disorder
* reaction to local anaesthetic
* infection
* any penile abnormality potentially complicating circumcision

Ages: 12 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Goldstuck, Study Director — University of Stellenbosch
Locations (1):
- Simunye Primary Healthcare, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Millard PS, Goldstuck ND. No-needle, single-visit adult male circumcision with Unicirc: a multi-centre field trial. PLoS One. 2015 Mar 30;10(3):e0121686. doi: 10.1371/journal.pone.0121686. eCollection 2015. PMID 25822727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unicirc Circumcision
Started | 54
Completed | 53
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Unicirc Circumcision
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Region of Enrollment [Number; unit: participants]
  South Africa | 54

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Duration
Description: Duration from placement of instrument to dressing
Time Frame: Intraoperative, 10-15 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Unicirc Circumcision
Number analyzed (Participants) | 54
minutes | 9.5 [9.5 to 10.0]

2. Secondary Outcome: Intraoperative Pain
Description: Intraoperative pain, measured on a standard 10 point pain scale (0=no pain, 5=moderate pain, 10 severe pain) using a pain face diagram.
Time Frame: Time of surgery, approximately 10-15 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale (0 - 10)
Arm/Group | Unicirc Circumcision
Number analyzed (Participants) | 54
units on a scale (0 - 10) | 1 [0.5 to 1.5]

3. Secondary Outcome: Healed at 4 Weeks
Description: Number of participants that are fully healed (epithelialized, no superficial ulcerations) at 4 weeks.
Time Frame: At the 4-week followup visit
Measure: Count of Participants; unit: Participants
Arm/Group | Unicirc Circumcision
Number analyzed (Participants) | 53
Participants | 53

ADVERSE EVENTS:
Time Frame: 1 month
Description: We looked for intra-operative or post-operative bleeding, hematoma, infection, poor cosmetic result, wound dehiscence. None of these or other events occurred.
Arm/Group | Unicirc Circumcision
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unicirc Circumcision (N=54)
Bleeding, hematoma, infection, wound dehiscence (Reproductive system and breast disorders) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no limitations, other than the fact that this study was not a comparison study but a cohort interventional study. Followup was not totally complete but very nearly so.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No